CLINICAL TRIAL: NCT01483976
Title: Comparison of Medical Nutritional Supplements With or Without AN777 in Elderly Men
Brief Title: Comparison of Medical Nutritional Supplements
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK96
Record Dates: First submitted 2011-11-23; First posted 2011-12-02 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral medical nutritional supplement without AN777 (Active Comparator): orally over a three hour period
  Interventions: Other: Oral medical nutritional supplement
- Experimental oral medical nutritional supplement with AN777 (Experimental): orally over a three hour period
  Interventions: Other: Experimental oral medical nutritional supplement with AN777

INTERVENTIONS:
Other: Oral medical nutritional supplement — orally over a three hour period
  Arms: Oral medical nutritional supplement without AN777
Other: Experimental oral medical nutritional supplement with AN777 — orally over a three hour period
  Arms: Experimental oral medical nutritional supplement with AN777

SUMMARY:
The objective of this study is to verify changes in protein metabolism after ingesting a oral medical nutritional supplement.

ELIGIBILITY:
Inclusion Criteria:

* Male and is ≥ 60 and ≤ 90 years of age.
* Body Mass Index (BMI) > 20.0, but < 35.0.
* Ability to climb a flight of 10 stairs or walk an equivalent of city block without help within the 3 months prior to enrollment.
* Refrain from taking any dose of NSAIDs or acetaminophen on the day of and 24 hours prior to Visit 2 and Visit 3.
* Refrain from using any pulmonary maintenance medications on the days of Visit 2 and Visit
* Refrain from intense physical activity between visits.

Exclusion Criteria:

* Systemic corticosteroids within the 3 months prior to enrollment.
* Blood thinner or anticoagulant medication within 1 week prior to enrollment.
* Glomerular filtration rate (eGFR) of < 40 mL/min/1.73m2.
* Antibiotics within 1 week prior to enrollment.
* Major surgery less than 3 months prior to enrollment in the study.
* Active malignant disease or treated within the last 6 months for cancer.
* Immunodeficiency disorder.
* Diabetes
* Myocardial infarction 3 months prior to enrollment.
* Chronic obstructive pulmonary disease
* History of allergy to any of the ingredients in the study products.
* Conditions precluding ingestion or absorption of the study product, inflammatory bowel disease, short bowel syndrome, or other major gastrointestinal disease.
* Dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder, or any other psychological condition.
* Pursuing weight loss or weight gain.
* Medications/dietary supplements/substances that could modulate metabolism or weight.

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in protein metabolism | Between baseline and 8 hours later
  Via amino acid tracers

SECONDARY OUTCOMES:
Intracellular signaling pathway metabolism | Between Baseline and 8 hours later
  Via Amino acid tracers and protein phosphorylation measurements

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States